CLINICAL TRIAL: NCT04738799
Title: The Impact of Food Order/Nutrient Sequence on Glycemic Excursions in Type 2 Diabetes Assessed by Continuous Glucose Monitoring
Brief Title: The Impact of Food Order on Glycemic Excursions in Type 2 Diabetes Assessed by Continuous Glucose Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20-03021613
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; nutrient sequence; food order; continuous glucose monitoring; cgm; t2dm; glycemic excursion; glp-1; ghrelin; insulin; cck; pyy; c-peptide; metformin; diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to continuous glucose monitoring readings.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate-Last Meal Sequence, Then Carbohydrate-First Meal Sequence (Experimental): Participants will consume the carbohydrate portion of their prepared meals last during mealtimes for 6 days. They will then consume the carbohydrate portion of their prepared meals first during mealtimes for the following 6 days.
  Interventions: Behavioral: Carbohydrate-Last Meal Sequence; Behavioral: Carbohydrate-First Meal Sequence
- Carbohydrate-First Meal Sequence, Then Carbohydrate-Last Meal Sequence (Experimental): Participants will consume the carbohydrate portion of their prepared meals first during mealtimes for 6 days. They will then consume the carbohydrate portion of their prepared meals last during mealtimes for the following 6 days.
  Interventions: Behavioral: Carbohydrate-Last Meal Sequence; Behavioral: Carbohydrate-First Meal Sequence

INTERVENTIONS:
Behavioral: Carbohydrate-Last Meal Sequence — Carbohydrates consumed last during mealtimes for 6 days
Behavioral: Carbohydrate-First Meal Sequence — Carbohydrates consumed first during mealtimes for 6 days

SUMMARY:
The purpose of this study is to explain the effect of food order/nutrient sequencing on glycemic excursions over a 2 week period, utilizing a device known as a continuous glucose monitor (CGM), for people who have been diagnosed with Type 2 Diabetes Mellitus and treated with metformin. This research study is being done because recent studies demonstrate that besides carbohydrate amount and type, the sequential order of macronutrient consumption during a meal has a significant impact on post-meal glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Metformin-treated type 2 diabetes of less than 10 years duration
* Must be on a stable dose of metformin for at least 1 month
* HbA1c ≤8.5 percent

Exclusion Criteria:

* Relevant food allergies
* Oral steroid therapy within 90 days of enrollment
* Anti-diabetic medications other than metformin
* History of bariatric surgery
* Pregnant women
* Any participant deemed unsuitable in the investigator's opinion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Change in incremental glucose peak, under controlled conditions | Day 6, Day 12
Change in mean amplitude of glycemic excursion, under controlled conditions | Day 6, Day 12
Change in time in range, under controlled conditions | Day 6, Day 12
  Time during which participant maintained a blood glucose level between 70-180mg/dL over 8 hour observation period

SECONDARY OUTCOMES:
Change in incremental glucose peak, under free-living conditions | Day 1 through 5, Day 7 through 11
Change in mean amplitude of glycemic excursion, under free-living conditions | Day 1 through 5, Day 7 through 11
Change in time in range, under free-living conditions | Day 1 through 5, Day 7 through 11
  Time during which participant maintained a blood glucose level between 70-180mg/dL
Change in postprandial insulin concentration | Day 6, Day 12
  Postprandial concentrations of insulin measured at 30-minute intervals for 180 minutes following standardized meal administration.
Change in postprandial c-peptide concentration | Day 6, Day 12
  Postprandial concentrations of c-peptide measured at 30-minute intervals for 180 minutes following standardized meal administration.
Change in postprandial ghrelin concentration | Day 6, Day 12
  Postprandial concentrations of ghrelin measured at 30-minute intervals for 180 minutes following standardized meal administration.
Change in postprandial PYY concentration | Day 6, Day 12
  Postprandial concentrations of PYY measured at 30-minute intervals for 180 minutes following standardized meal administration.
Change in postprandial GLP-1 concentration | Day 6, Day 12
  Postprandial concentrations GLP-1 measured at 30-minute intervals for 180 minutes following standardized meal administration.
Change in postprandial CCK concentration | Day 6, Day 12
  Postprandial concentrations of CCK measured at 30-minute intervals for 180 minutes following standardized meal administration.
Change in satiety, as measured by Visual Analog Scale (VAS) | Day 6, Day 12
  Scores are measured on a 100mm VAS. The VAS ranges from 0 to 100, with 0 indicating lower satiety and higher scores indicating greater satiety.

CONTACTS AND LOCATIONS:
Overall Officials: Alpana Shukla, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No